CLINICAL TRIAL: NCT00443625
Title: Clinical Trials to Investigate the Influence of Food on Pharmacokinetics of SK3530 in Healthy Male Volunteers.
Brief Title: Phase 1 Study of SK3530 to Investigate of the Effect of Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SK3530_FE
Record Dates: First submitted 2007-02-22; First posted 2007-03-06 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Erectile Dysfunction
Keywords: SK3530; Food effect; Pharmacokinetics
MeSH Terms: conditions — Erectile Dysfunction | interventions — 2-(5-(4-(2-hydroxyethyl)piperazin-1-ylsulfonyl)-2-n-propoxyphenyl)-5-ethyl-7-n-propyl-3,5-dihydro-4H-pyrrolo(3,2-d)pyrimidin-4-one dihydrochloride

INTERVENTIONS:
Drug: SK3530

SUMMARY:
This study was designed to investigate the food effect of SK3530 on the pharmacokinetics (PKs).

DETAILED DESCRIPTION:
The PDE5 inhibitor, SK3530, is expected to be taken concomitantly with food. The food interaction studies of other PDE5 inhibitors (Viagra, Levitra and cialis) have already accomplished and the results have provided useful information to the patients. The objective of this study is to compare the pharmacokinetics (PKs) of SK3530 and its metabolite (SK3541) under the fasted and fed (low-fat meal and high-fat meal) conditions.

ELIGIBILITY:
Inclusion Criteria:

* ages 19 to 50
* body weight of (IBM) ± 20%

Exclusion Criteria:

* cardiovascular disease
* color-blindness or weakness

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15
Dates: Start 2006-12; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
PK parameters - AUC, Cmax, Tmax

SECONDARY OUTCOMES:
PK parameters-t1/2

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, Principal Investigator — Seoul National University Hospital